CLINICAL TRIAL: NCT01926652
Title: An Open-label, Multiple-dosing, Two-arm, One-sequence, Crossover Study to Evaluate the Safety and Pharmacokinetics After Oral Concurrent Administration of Amlodipine 10mg and Candesartan 32mg in Healthy Male Volunteers
Brief Title: Safety and Pharmacokinetics Study of Amlodipine 10mg and Candesartan 32mg
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shin Poong Pharmaceutical Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: SP-AC-001
Record Dates: First submitted 2013-08-18; First posted 2013-08-21 (Estimated); Last update posted 2013-08-21 (Estimated); Status verified 2013-08

CONDITIONS: Healthy
MeSH Terms: interventions — candesartan cilexetil; Amlodipine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- candesartan (Experimental): Single administration : candesartan cilexetil 32mg, qd. Combination administration : candesartan cilexetil 32mg and amlodipine 10mg, qd
  Interventions: Drug: candesartan cilexetil 32mg, amlodipine 10mg
- amlodipine (Experimental): Single administration : amlodipine 10mg, qd. Combination administration : candesartan cilexetil 32mg and amlodipine 10mg, qd
  Interventions: Drug: candesartan cilexetil 32mg, amlodipine 10mg

INTERVENTIONS:
Drug: candesartan cilexetil 32mg, amlodipine 10mg — Part A: Treatment A (candesartan), Treatment B (candesartan + amlodipine) 2-period, 2-treatment crossover.
  Part B: Treatment A (Amlodipine), Treatment B (candesartan + amlodipine) 2-period, 2-treatment crossover.
  Other Names: atacand 32mg, norvasc 10mg

SUMMARY:
Clinical trial to evaluate the pharmacokinetic interactions and safety between single dose of amlodipine 10mg and candesartan 32mg and the combination dose amlodipine 10mg with candesartan 32mg in healthy male volunteers.

ELIGIBILITY:
Inclusion Criteria:

1. Male volunteers in the age between 20 and 55 years old(inclusive).
2. Body weight >= 55kg and Body mass index (BMI) in the range of calculated IBW ±20%.
3. Subjects without a hereditary problems or chronic desease.
4. Subjects whose clinical laboratory test values are inside the accepted normal range.
5. Understand the requirements of the study and voluntarily consent to participate in the study.

Exclusion Criteria:

1. Subjects with a history of gastrointestinal diseases which might significantly change ADME of medicines.
2. Systolic blood pressure range ≥150 mmHg or ≤ 100 mmHg or diastolic blood pressure range ≥ 95 mmHg or ≤ 60 mmHg.
3. Subject with symptoms of acute disease within 14days prior to study medication dosing.
4. Subjects with a history of clinically significant allergies of amlodipin or candesartan or CCB or other medicine (ex. aspirin or antibiotics).
5. Subjects with galactose intolerance, Lapp lactase deficiency or glucose-galactose malabsorption.
6. Serum creatinine > 1.2mg/dL.
7. smoking > 10 cigarettes/day.
8. alcohol > 210g/week.
9. Positive test results for drug test in urin or subject with history of substance abuse.
10. Participation in any clinical investigation within 2 months prior to study medication dosing.
11. Subjects with whole blood donation within 2 months, component blood donation within 1 month and blood transfusion within 1 month prior to study medication dosing.
12. Subjects considered as unsuitable based on medical judgement by investigators.

Ages: 20 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2013-07; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
AUC, Cmax | 7days, 10days

SECONDARY OUTCOMES:
Cmin, tmax, CL/F | 7days, 10days

CONTACTS AND LOCATIONS:
Locations (1):
- Chungnam national university hospital, clinical trial center, Daejeon, Chungcheongbul-do, South Korea